CLINICAL TRIAL: NCT04526197
Title: A Phase 1, Randomized, 2-Period, 2-Sequence, Cross-over Study to Determine the Effect of ALXN1840 on the Metabolism of a CYP2C9 Substrate in Healthy Participants.
Brief Title: Phase 1 Study of ALXN1840 on the Metabolism of a CYP2C9 Substrate in Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1840-HV-105
Record Dates: First submitted 2020-08-19; First posted 2020-08-25 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2022-10

CONDITIONS: Wilson Disease
Keywords: Cytochrome P450; Healthy; ALXN1840; Celecoxib; CYP2C9
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — tetrathiomolybdate; Celecoxib

STUDY DESIGN:
Intervention Model Description: Participants were randomized to 1 of 2 treatment sequences: A-B or B-A.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence A-B (Experimental): Participants received 1 treatment during each study period in the following sequence:
  * Treatment A: Celecoxib.
  * Treatment B: Celecoxib plus ALXN1840.
  Interventions: Drug: ALXN1840; Drug: Celecoxib
- Treatment Sequence B-A (Experimental): Participants received 1 treatment during each study period in the following sequence:
  * Treatment B: Celecoxib plus ALXN1840.
  * Treatment A: Celecoxib.
  Interventions: Drug: ALXN1840; Drug: Celecoxib

INTERVENTIONS:
Drug: ALXN1840 — ALXN1840 was administered orally as a single dose as 4 x 15 milligram (mg) enteric-coated tablets with 240 milliliters (mL) of water (fasting), for a total dose of 60 mg.
  Other Names: WTX101; Bis-choline tetrathiomolybdate; Tiomolibdate choline
Drug: Celecoxib — Celecoxib was administered orally as a single dose as one 200-mg tablet with 240 mL of water (fasting).

SUMMARY:
This was a Phase 1, randomized, 2-period, 2-sequence, cross-over study designed to determine the effect of ALXN1840 on the metabolism of celecoxib, a sensitive cytochrome P450 2C9 (CYP2C9) substrate, in healthy male and female participants. The safety and tolerability of ALXN1840 were determined along with ALXN1840 pharmacokinetics (PK) in plasma as measured via total molybdenum with the coadministration of celecoxib.

DETAILED DESCRIPTION:
The study was conducted as a randomized, 2-period, 2-sequence, cross-over study to determine the effect of a single dose of ALXN1840 (perpetrator) on the single-dose celecoxib (victim) kinetics in healthy male and female participants.

The study had a Screening period (Day -28 to Day -2), two 11-day study periods (Day 1 to Day 11) with a minimum of 14 days between doses of celecoxib, and an End of Study Visit (Day 15 ± 2 days) after Period 2 dosing. Participants only reported to the clinical research unit (CRU) on the day prior to the first dose because they were kept in the CRU during the wash-out period due to coronavirus disease 2019.

All participants received a single dose of celecoxib alone (Treatment A) and celecoxib coadministered with ALXN1840 (Treatment B) during the study, 1 in each treatment period. Based on randomization, participants were administered either Treatments A-B or Treatments B-A in each study period.

The PK profile of ALXN1840 and celecoxib was determined by blood sampling following single-dose administration. In addition to PK sampling, safety and tolerability were assessed by monitoring adverse events, vital signs, 12-lead electrocardiograms, physical examinations, and laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adequate venous access in the left or right arm to allow the collection of blood samples.
* Bodyweight ≥ 45 to ≤ 100 kilograms (kg) and body mass index within the range of 18 to < 30 kg/meter squared.
* Willing and able to follow protocol-specified contraception requirements.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of/significant medical history.
* Clinically significant multiple or severe allergies.
* Lymphoma, leukemia, or any malignancy within 5 years.
* Breast cancer within the past 10 years.
* Serum creatinine > upper limit of normal (ULN) of the reference range.
* Alanine aminotransferase, aspartate aminotransferase, or total bilirubin > ULN.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QTc > 450 milliseconds (msec) for male participants or > 470 msec for female participants.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 70 potential participants were screened for this study, and 36 participants were randomized.
Pre-assignment Details: Participants were randomized to 1 of 2 treatment sequences (A-B) or (B-A) in a crossover study design during 2 dosing periods. Participants were scheduled to receive either treatment A or B on Day 1 of each dosing period. There was a washout of at least 14 days between the dosing periods.
Groups:
- Treatment Sequence A-B; Treatment Sequence B-A: All participants were randomized to 1 of 2 treatment sequences (A-B or B-A) and received 1 treatment in each study period; treatment order was defined based on randomization:
  * Treatment A: Celecoxib.
  * Treatment B: Celecoxib plus ALXN1840.
Period: Period 1
Arm/Group | Treatment Sequence A-B | Treatment Sequence B-A
Started | 18 | 18
Received at Least 1 Dose of Study Drug | 18 | 18
Completed | 17 | 17
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 2
Arm/Group | Treatment Sequence A-B | Treatment Sequence B-A
Started | 17 | 17
Received at Least 1 Dose of Study Drug | 17 | 17
Completed | 17 | 15
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug during treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence A-B | Treatment Sequence B-A | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.5 (8.79) | 33.9 (7.01) | 34.2 (7.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 13 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 6 | 17
  Not Hispanic or Latino | 7 | 12 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Black or African American | 4 | 7 | 11
  White | 13 | 11 | 24
Height [Mean (Standard Deviation); unit: Centimeters] | 170.61 (8.225) | 168.21 (6.997) | 169.41 (7.624)
Weight [Mean (Standard Deviation); unit: Kilograms] | 77.29 (10.466) | 72.06 (9.886) | 74.67 (10.378)
Body Mass Index [Mean (Standard Deviation); unit: Kilograms/squared meter] | 26.43 (1.856) | 25.41 (2.596) | 25.92 (2.283)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) Of Celecoxib With And Without The Coadministration Of ALXN1840
Description: Blood samples were collected for pharmacokinetics (PK) analysis of celecoxib. Cmax is reported as nanograms (ng)/milliliter (mL).
Time Frame: Baseline, up to 336 hours post-dose
Population: Pharmacokinetic Analysis Set: All randomized participants who received both study drugs and had sufficient plasma samples for evaluable PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Treatment A: Participants who received celecoxib.
- Treatment B: Participants who received celecoxib with ALXN1840.
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 35 | 35
ng/mL | 637.1 (48.7) | 567.4 (49.4)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Other — Confidence Interval; Ratio of geometric LS means = 0.881, 90% CI 2-sided [0.776 to 1.001]

2. Primary Outcome: Area Under The Plasma Concentration Versus Time Curve From Time 0 To The Last Quantifiable Concentration (AUCt) Of Celecoxib With And Without The Coadministration Of ALXN1840
Description: Blood samples were collected for pharmacokinetic (PK) analysis of celecoxib. Area Under The Plasma Concentration Versus Time Curve From Time 0 To The Last Quantifiable Concentration (AUCt) is reported as hours•ng/mL (h•ng/mL).
Time Frame: Baseline, up to 336 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h•ng/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 35 | 35
h•ng/mL | 6406 (40.8) | 6482 (39.9)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Other — Confidence Interval; Ratio of geometric LS means = 1.016, 90% CI 2-sided [0.959 to 1.077]

3. Primary Outcome: Area Under The Plasma Concentration Versus Time Curve From Time 0 To Infinity (AUCinf) Of Celecoxib With And Without The Coadministration Of ALXN1840
Description: Blood samples were collected for pharmacokinetic (PK) analysis of celecoxib. Area Under The Plasma Concentration Versus Time Curve From Time 0 To Infinity (AUCinf) is reported as h•ng/mL.
Time Frame: Baseline, up to 336 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h•ng/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 35 | 35
h•ng/mL | 6743 (38) | 6869 (37.8)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Other — Confidence Interval; Ratio of geometric LS means = 1.010, 90% CI 2-sided [0.954 to 1.070]

4. Secondary Outcome: Cmax Of Molybdenum With Coadministration Of Celecoxib
Description: Blood samples were collected for PK analysis of total molybdenum (as a measure of ALXN1840) and plasma ultrafiltrate (PUF) molybdenum. Cmax is reported as ng/mL.
Time Frame: Baseline, up to 336 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment B
Number analyzed (Participants) | 35
ng/mL
  Total Molybdenum | 373.4 (44.8)
  PUF Molybdenum | 82.44 (75.5)

5. Secondary Outcome: AUCt Of Molybdenum With Coadministration Of Celecoxib
Description: Blood samples were collected for PK analysis of total molybdenum (as a measure of ALXN1840) and PUF molybdenum. AUCt is reported as h•ng/mL.
Time Frame: Baseline, up to 336 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h•ng/mL
Arm/Group | Treatment B
Number analyzed (Participants) | 35
h•ng/mL
  Total Molybdenum | 19240 (49.1)
  PUF Molybdenum | 1796 (50.8)

6. Secondary Outcome: AUCinf Of Molybdenum With Coadministration Of Celecoxib
Description: Blood samples were collected for PK analysis of total molybdenum (as a measure of ALXN1840) and PUF molybdenum. AUCinf is reported as h•ng/mL.
Time Frame: Baseline, up to 336 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h•ng/mL
Arm/Group | Treatment B
Number analyzed (Participants) | 35
h•ng/mL
  Total Molybdenum: number analyzed (Participants) | 33
  Total Molybdenum | 20910 (47.3)
  PUF Molybdenum: number analyzed (Participants) | 8
  PUF Molybdenum | 2305 (36.5)

ADVERSE EVENTS:
Time Frame: Day 1 through 15 (± 2) days after final dose of study drug.
Arm/Group | Treatment A | Treatment B
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 8/35 | 3/35
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=35) | Treatment B (N=35)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dental discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT04526197/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT04526197/SAP_001.pdf